CLINICAL TRIAL: NCT04830215
Title: A Phase 4, Multicenter, Open-label, Interventional Trial to Assess the Effects on Engagement of Flexible-dose Brexpiprazole (OPC-34712) as Adjunctive Therapy for the Treatment of Adults With Major Depressive Disorder
Brief Title: Brexpiprazole as Adjunctive Therapy in Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Lundbeck Canada Inc. (Industry); Otsuka Canada Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-201-00289
Record Dates: First submitted 2021-03-29; First posted 2021-04-05 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-05

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Depression; Brexpiprazole
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brexpiprazole (Other): Participants received brexpiprazole as a flexible dose; 0.5 mg to 2 mg, orally (PO), QD, and continued on the stable dose of ADT up to 8 weeks.
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Oral brexpiprazole tablets as adjunctive therapy to ADT
  Other Names: OPC-34712

SUMMARY:
The clinical trial will investigate the effect of brexpiprazole on the concept of life engagement in participants with Major Depressive Disorder (MDD) with a current depressive episode.

DETAILED DESCRIPTION:
This is a phase 4, multicenter, open-label, flexible dose trial designed to assess the effects of brexpiprazole (flexible dose; 0.5 to 2 milligrams [mg], once daily [QD]) as adjunctive therapy to antidepressant therapy (ADT) on life engagement in participants with MDD. This trial is being conducted in line with the Canadian Product Monograph.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants (outpatients) between the regional age of majority (18 or 19 years of age) to 65 years of age, inclusive, at the time of informed consent.
* Primary diagnosis of MDD and in a current non-psychotic major depressive episode (MDE) as defined by Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria, who have been outpatients for at least 4 weeks, and have an inadequate response, per investigator judgment, to 1 or 2 adequate treatments of ADTs in their current MDE, including current ADT.
* Participants with a Patient Health Questionnaire 9-item scale (PHQ-9) ≥ 15 at the screening and baseline visits, if separate.

Exclusion Criteria:

* Participants currently or previously treated with brexpiprazole including participants who received brexpiprazole in any prior clinical trial.
* Participants with a concurrent DSM-5 diagnosis of the following will be excluded:

  * Schizophrenia or schizoaffective disorder
  * Bipolar I or bipolar II disorder
  * Post-traumatic stress disorder
  * Dementia
  * Eating disorder
  * Borderline personality disorder
  * Antisocial personality disorder
* Participants with a suicidality score of 3 based on Inventory of Depressive Symptomatology Self-Report (IDS-SR) suicidality item 18 or participants who, in the opinion of the investigator, presents a serious risk of suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (1):
- Chatham-Kent Clinical Trials Research Centre, Chatham, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Therrien F, Chokka P, Habert J, Ismail Z, McIntyre RS, Dine J, Brown TM, Zhang Z, MacKenzie EM, Ward CL. Patient-reported efficacy of adjunctive brexpiprazole in major depressive disorder in a phase 4, open-label, interventional study. Curr Med Res Opin. 2025 Aug;41(8):1511-1522. doi: 10.1080/03007995.2025.2558140. Epub 2025 Sep 16. PMID 40913583
- [Derived] Therrien F, Ward C, Chokka P, Habert J, Ismail Z, McIntyre RS, MacKenzie EM. Adjunctive Brexpiprazole for Patient Life Engagement in Major Depressive Disorder: A Canadian, Phase 4, Open-Label, Interventional Study: Brexpiprazole d'appoint pour l'engagement dans la vie des patients souffrant de trouble depressif majeur: une etude interventionnelle canadienne ouverte de phase 4. Can J Psychiatry. 2024 Jul;69(7):513-523. doi: 10.1177/07067437241233965. Epub 2024 Mar 1. PMID 38425284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 15 investigative sites in Canada from 01 April 2021 to 27 May 2022.
Pre-assignment Details: A total of 157 participants were screened of which 122 participants were enrolled and 120 participants were treated in the study.
Groups:
- Brexpiprazole: Participants received brexpiprazole as a flexible dose; 0.5 milligrams (mg) to 2 mg, orally (PO), once daily (QD), and continued on the stable dose of antidepressant therapy (ADT) up to 8 weeks.
Period: Overall Study
Arm/Group | Brexpiprazole
Started | 122
Efficacy Analysis Set (The Efficacy Analysis Set included all participants who had a baseline value and at least one post-baseline efficacy evaluation for Inventory of Depressive Symptomatology Self-Report (IDS-SR) total score and IDS-SR-10-engagement during the open label treatment phase.) | 120
Safety Analysis Set (The Safety Analysis Set included all participants who received at least one dose of open-label brexpiprazole.) | 120
Completed | 111
Not Completed | 11
Not completed — Adverse Event | 6
Not completed — Failure to Meet Continuation Criteria | 1
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Deviation | 1

BASELINE CHARACTERISTICS:
Population: The Enrolled Analysis Set included all participants who had signed the informed consent form (ICF) for the trial and had enrolled into the open-label treatment phase.
Groups:
- Brexpiprazole: Participants received brexpiprazole as a flexible dose; 0.5 mg to 2 mg, PO, QD, and continued on the stable dose of ADT up to 8 weeks.
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 111
  Race: Black or African American | 1
  Race: Asian | 7
  Race: Other | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1
  Ethnicity: Not Hispanic or Latino | 117
  Ethnicity: Unknown | 3
  Ethnicity: Other | 1
IDS-SR-10 Engagement [Mean (Standard Deviation); unit: score on a scale] — Population: Efficacy Analysis Set included all participants who had a baseline value and at least one post-baseline efficacy evaluation for IDS-SR total score and IDS-SR-10 engagement during the open label treatment phase. IDS-SR-10-engagement consist of selected 10 item scores, including the following 10 items (clinician-selected): items 8, 15, 16, 17, 19, 20, 21, 22, 23, and 29. All 10 items are rated on a 0 (best) to 3 (worst) scale. The total score ranges from 0 (best) to 30 (worst).
  score on a scale
    number analyzed (Participants) | 120
    (all) | 16.1 (4.7)
IDS-SR Total Score [Mean (Standard Deviation); unit: score on a scale] — Population: Efficacy Analysis Set. IDS-SR is 30-item self-report measure used to assess core diagnostic depressive symptoms & atypical & melancholic symptom features of major depressive disorder(MDD).Each item rated=0(best)-3(worst).It is sum of ratings of 28 items. Total score=0(best)-84(worst).Item 9 has 2 subitems 9A (score=1,2,&3)& 9B (score=0 or 1).Scores for 9A & 9B are not included in calculation of total score.Item 11/12 should be completed but not both, item 13/14 should be completed but not both.
  score on a scale
    number analyzed (Participants) | 120
    (all) | 41.3 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in IDS-SR-10 Engagement
Description: The IDS-SR-10 engagement consist of selected 10 item scores, including the following 10 items (clinician-selected): item 8 - Response of your mood to good or desired events, item 15 - Concentration/decision making, item 16 - View of myself, item 17 - View of my future, item 19 - General interest, item 20 - Energy level, item 21 - Capacity for pleasure or enjoyment (excluding sex), item 22 - Interest in sex (interest rated, not activity), item 23 - Feeling slowed down, and item 29- Interpersonal sensitivity. All the 10 items are rated on a 0 (best) to 3 (worst) scale. IDS-SR-10 engagement total score ranges from 0 (best) to 30 (worst). A negative change from baseline indicated improvement. Least square (LS) mean was calculated using a mixed model repeated measure (MMRM) analysis.
Time Frame: Baseline to Week 8
Population: The Efficacy Analysis Set included all participants who had a baseline value and at least one post-baseline efficacy evaluation for IDS-SR total score and IDS-SR-10-engagement during the open label treatment phase. Overall number analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 105
score on a scale | -8.11 (0.62)
Statistical Analysis 1: Comparison: Brexpiprazole; Test type: Other; p < 0.0001, MMRM — MMRM included fixed effect terms for visit, baseline value, an interaction term of baseline value by visit, and trial center

2. Primary Outcome: Change From Baseline in IDS-SR Total Score
Description: The IDS-SR is a 30-item self-report measure that was used to assess core diagnostic depressive symptoms as well as atypical and melancholic symptom features of major depressive disorder (MDD). Each item on the IDS-SR scale was rated on a 0 to 3 scale with 0 being the "best" rating and 3 being the "worst" rating. IDS-SR total score is the sum of ratings of 28 item scores with the total score ranging from 0 (best) to 84 (worst). Under item 9, two sub-items 9A and 9B exist, with possible scores of 1, 2 or 3 for item 9A, and 0 or 1 for item 9B. The scores for these two sub-items are not included in the calculation of the total score. Item 11 or item 12 should be completed but not both, and similarly, item 13 or item 14 should be completed but not both. A negative change from baseline indicated improvement. LS mean was calculated using a MMRM analysis.
Time Frame: Baseline to Week 8
Population: The Efficacy Analysis included all participants who had a baseline value and at least one post-baseline efficacy evaluation for IDS-SR total score and IDS-SR-10-engagement during the open label treatment phase. Overall number analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole
Number analyzed (Participants) | 105
score on a scale | -17.38 (1.36)
Statistical Analysis 1: Comparison: Brexpiprazole; Test type: Other; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 8
Description: The Safety Analysis Set included all participants who received at least one dose of open-label brexpiprazole.
Arm/Group | Brexpiprazole
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 45/120
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=120)
Nausea (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 13
Weight increased (Investigations) | 7
Headache (Nervous system disorders) | 13
Tremor (Nervous system disorders) | 8
Insomnia (Psychiatric disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT04830215/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT04830215/SAP_001.pdf